CLINICAL TRIAL: NCT03005444
Title: Anticoagulation for Development of Further Decompensation and Survival in Advanced Cirrhosis After Transjugular Intrahepatic Portosystemic Shunt: a Multicenter Randomized Controlled Study
Brief Title: Anticoagulation for Advanced Cirrhotic Patients After TIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, MD，PhD，Professor, Xi'an International Medical Center Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APPROACH
Record Dates: First submitted 2016-12-21; First posted 2016-12-29 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; Transjugular Intrahepatic Portosystemic Stent Shunt; Anticoagulation; Survival; Additional decompensation
MeSH Terms: conditions — Liver Cirrhosis | interventions — Rivaroxaban; Nadroparin; Enoxaparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anticoagulation (Experimental): Rivaroxaban：10mg/d for 2 years
  Interventions: Drug: Rivaroxaban
- Non-anticoagulated (No Intervention): No anticoagulants will be used.

INTERVENTIONS:
Drug: Rivaroxaban — 10mg/day, for 2 years
  Other Names: Nadroparin or Enoxaparin
  Arms: Anticoagulation

SUMMARY:
Recent studies demonstrated that liver cirrhosis was associated with a hypercoagulability state. Besides, bacterial translocation plays an important role in the pathogenesis and complications in patients with decompensated cirrhosis, including infections as well as hepatic encephalopathy and hepatorenal syndrome.

A recent prospective study in a group of 70 patients with liver cirrhosis (Child B and C stages up to 10 points) who were randomized to receive enoxaparin for a year (n = 34) vs no intervention (n = 36) showed that anticoagulant treatment with enoxaparin is safe and effective, significantly reducing risk of PVT development and liver decompensation, markedly improving overall survival. This study provides exciting preliminary data regarding the potential use of prophylactic anticoagulation in improving clinical outcomes in cirrhosis, beyond the prevention of portal vein thrombosis. This study suggested that the effect was partly due to a direct effect of reducing BT and levels of proinflammatory cytokines. However, this study included few patients, was not double blind, and did not have a placebo group. Therefore, despite the spectacular results, the use of prophylactic anticoagulant therapy has not become routine practice in patients with cirrhosis and more studies are needed to assess the potential usefulness of anticoagulation in improving the prognosis of liver cirrhosis.

Transjugular intrahepatic portosystemic shunts (TIPS) are now routinely used to treat the complications of portal hypertension, such as variceal bleeding and refractory ascites. TIPS is the most effective method to prevent rebleeding, however, it is burdened with increased risk of hepatic encephalopathy and deterioration of liver function in patients with advanced cirrhosis. Notably, TIPS can not only relieve portal pressure but also can redirect the portal blood flow through the shunt directly into the systemic circulation which can cause systemic hemodynamic changes.

Given the preliminary data suggesting a beneficial effect of prophylactic anticoagulation with LMWH in cirrhotic patients, this multicenter randomized controlled study attempts to demonstrate the effect of long term LMWH therapy after TIPS on survival in cirrhotic patients with variceal bleeding.

ELIGIBILITY:
All inclusion criteria must be met at the time of screening:

* Signed informed consent.
* Male or female patients with an age of 18 to 75 years
* Liver cirrhosis.
* History of variceal bleeding > 5 days
* Presence of ascites
* Successful TIPS
* Use of Viatorr stent
* Child-Pugh score within B7-C13
* Bilirubin level of 3 mg/dL or less (51.3 umol/L)

Patients who meet the following criteria at the time of screening will be excluded:

* Hepatocellular carcinoma or other intrahepatic/extrahepatic cancers.
* Spontaneous overt hepatic encephalopathy.
* Previous or current portal venous system thrombosis.
* Budd-Chiari syndrome.
* Known coagulation disorder besides liver cirrhosis.
* Severe thrombocytopenia <15,000 platelets/dl.
* Peptic ulcer disease in the last 6 months.
* Unstable angina or myocardial infarction (MI) within the past 6 months before randomization.
* Cardiac arrhythmias requiring anti-arrhythmic therapy (beta blockers or digoxin are permitted).
* Uncontrolled hypertension.
* Prior liver transplantation or candidates for liver transplantation.
* History of shunting surgery or TIPS before randomization.
* Pregnancy or breastfeeding
* Poor compliance
* Participation in another clinical trial
* Close affiliation with the investigational site.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival | 2 years

SECONDARY OUTCOMES:
Number of participants with all-cause rebleeding | 2 years
Number of participants with overt hepatic encephalopathy | 2 years
Number of participants with recurrent or worsening ascites | 2 years
  Perform two or more evacuative paracentesis in the following six months
Number of participants with shunt dysfunction | 2 years
Effect of anticoagulation on liver function estimated by the Child-Pugh and the model for end-stage liver disease scores | 2 years
Echocardiography findings | 2 years
Serum levels of bacterial translocation biomarkers and proinflammatory cytokines | 2 years
Security of anticoagulation in patients with liver cirrhosis | 2 years
  Number of adverse events and adverse reactions in each arm of study. History and clinical evaluation of bleeding and monitoring of hematocrit.
Compliance | 2 years
  Record of unused packaging and information about compliance in a patient diary
Score of Health Related Quality of Life questionnaire，for example, SF-36 | 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital Affiliated to Southern Medical University, Guanzhou, Guangdong
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The first affiliated hospital of Nanchang university, Nanchang, Jiangxi
  - The First Affiliated Hospital, Air Force Medical University, Xi'an, Shaanxi
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Provincial Hospital Affiliated to Shandong University, Jinan, Shandong
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang